CLINICAL TRIAL: NCT01908114
Title: To Develop, Implement and Evaluate the Polio Demonstration Project Comprising of a Community Based Intervention Package for Polio Eradication in Pakistan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Pakistan Ministry of Health (Other Government); Trust for Vaccines and Immunization, Pakistan (Other); National Institutes of Health, Pakistan (Other); Peshawar Medical College (Other); World Health Organization (Other); UNICEF (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Founding Director, Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2432-PED-ERC-12
Record Dates: First submitted 2013-07-15; First posted 2013-07-25 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Polio; Polio Sero Conversion; Polio Sero Prevalence; Immunization Coverage
Keywords: Polio disease; Intervention Package; Polio sero prevalence and sero conversion; Polio high risk areas of Pakistan
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (No Intervention): Routine Polio Program activities will be carried out with out any active intervention
- Group B (Experimental): Expanded intervention with following components
  1. Community support groups for both male and female at village/community level
  2. Enhanced communication package and involvement of local social networks for group counseling on promotion of nutrition, hygiene and Expanded Program of Immunization (EPI) vaccinations
  3. Involvement of Private sector (General Physicians,health care providers etc.) through advocacy and inclusion in Supplementary Immunization activities (SIAs)
  4. Delivery of interventions & commodities through low cost health camps during National Immunization days (NIDs) and SIAs (will also assist in mop-up campaigns)
  Interventions: Behavioral: Enhanced Community mobilization
- Group C (Experimental): All Interventions of Group A and B Plus combined bOPV/IPV strategy in the SIAs during the project
  Interventions: Behavioral: Enhanced Community mobilization; Biological: Combined Oral Polio Vaccine and Inject able Polio Vaccine during SIA

INTERVENTIONS:
Behavioral: Enhanced Community mobilization
  Arms: Group B; Group C
Biological: Combined Oral Polio Vaccine and Inject able Polio Vaccine during SIA
  Arms: Group C

SUMMARY:
The objective of the projects is to Develop and implement a Package of interventions that will comprise of an augmented communication and counseling strategy coupled with private sector involvement and a combined Oral Polio Vaccine and Inject able Polio Vaccine approach during the Polio campaigns followed by the evaluation of this project for acceptability, feasibility and effectiveness of the intervention Package.

DETAILED DESCRIPTION:
This particular project has been designed to address the bottlenecks through innovations to address community mobilization and demand creation on one hand and assess the synergistic immune enhancement potential of combining Inject able Polio Vaccine (IPV) and Oral Polio Vaccine (OPV) in at-risk children. This project will be implemented in high risk union councils of Karachi, district Kashmore in Sindh and Bajaur Agency in Federally administered Tribal areas (FATA)

This will be a three cell cluster randomized trial to achieve the objectives of the study. The first cell of the study will receive all the routine activities being carried out by the polio program, the second cell will receive an expanded intervention with community support groups, enhanced communication package, education and counseling and involvement of private sector. While the third cell will receive all of the interventions of second cell with a combined OPV IPV approach during the polio immunization campaign through child health camps.

We have calculated a total sample size of 120 clusters, 40 clusters per group for each study area i-e 120 for Karachi, 120 for Kashmore and 120 for Bajaur. Polio program in Pakistan has well established and demarcated vaccination areas assigned to a vaccination team, each vaccination area usually covers about 200 children therefore the area of vaccination team will be considered as one cluster in the proposed study.

The implementation of the project will be followed by impact assessment activities that will include post vaccination coverage surveys and Immunity assessment activities and Environmental sample collection. A total sample size of 5310 children has been calculated for the immunity studies for seroprevalance and 5130 for stool virus shedding

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 1 month to 5 years that reside within the study sites, and do not plan to travel away during entire the study period.

Exclusion Criteria:

* Children with known thrombocytopenia or bleeding disorders; children acutely ill or with signs of acute infection (e.g. fever ≥ 101 F) at the time of NID and a diagnosis or suspicion of immunodeficiency disorder.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60000 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improved immunization coverage | At the completion of all recruitment and follow ups which will take an average time of 1 year
  Improved coverage in both routine immunization and polio campaign Immunization compared to Baseline

SECONDARY OUTCOMES:
Improved Polio Sero prevalence | The immunity levels will be assessed at the time of recruitment, six weeks after recruitment and 18 weeks after recruitment
  Population bases Immunity level for polio antibodies will be assessed by
  Sero prevalance and conversion at various time points
Quantification of Polio virus in stool samples | The stool samples will be collected and analysed at day 28, day 35 and day 49 after recruitment
  Quantification of Polio virus will be assessed in stool samples collected at day 28, day 35 and day 49 after recruitment
Shedding of Polio virus in stool samples | The stool samples will be collected and analysed at day 28, day 35 and day 49 after recruitment
  Shedding of Polio virus in stool samples will be assessed at day day 28, day 35 and day 49 after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Habib MA, Soofi S, Cousens S, Anwar S, Haque NU, Ahmed I, Ali N, Tahir R, Bhutta ZA. Community engagement and integrated health and polio immunisation campaigns in conflict-affected areas of Pakistan: a cluster randomised controlled trial. Lancet Glob Health. 2017 Jun;5(6):e593-e603. doi: 10.1016/S2214-109X(17)30184-5. PMID 28495264